CLINICAL TRIAL: NCT02931799
Title: Prevention of Readmissions at Inflammatory Bowel Disease Centres of Excellence
Brief Title: Prevention of Readmissions at IBD Centres of Excellence
Acronym: PRICE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Crohn's and Colitis Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PRICE
Record Dates: First submitted 2016-10-11; First posted 2016-10-13 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Colitis, Ulcerative; Crohn Disease; Inflammatory Bowel Diseases
Keywords: Colitis, Ulcerative; Crohn Disease; Inflammatory Bowel Diseases; Gastroenterology; Quality Improvement; Post-Discharge
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Inflammatory Bowel Diseases | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse Follow-Up and Electronic Monitoring (Experimental)
  Interventions: Behavioral: Nurse Follow-Up; Other: Electronic Monitoring; Other: Post-Discharge Questionnaire; Other: Standard of Care
- Minimal Intervention (Active Comparator)
  Interventions: Other: Post-Discharge Questionnaire; Other: Standard of Care

INTERVENTIONS:
Behavioral: Nurse Follow-Up — Organized follow-up with an IBD advanced practice nurse at 24-48 hours, 7 days, and 30 days post-discharge; to monitor patients' health status with respect to their IBD.
  Arms: Nurse Follow-Up and Electronic Monitoring
Other: Electronic Monitoring — Patients will be provided access to a web-based application entitled: 'Health Promise'. The application will generate surveys every 3 days, where patients will self-report their IBD symptoms, quality of life and medication adherence on three separate scales:
  * PRO-2 Scale for patients with Crohn's Disease
  * 6-Point Mayo Score for patients with Ulcerative Colitis
  * Morisky Medication Adherence Scale (MMAS-4)
  The survey responses will be monitored by an IBD advanced practice nurse, to triage patients for outpatient follow-up.
  Arms: Nurse Follow-Up and Electronic Monitoring
Other: Post-Discharge Questionnaire — Patients will complete a web-based questionnaire at 30 days post-discharge. The questionnaire will capture information related to: Demographics, Patient Satisfaction as measured by the CACHE questionnaire; IBD related quality of life as measured by the IBDQ questionnaire; Disease activity as measured by PRO-2 scale for Crohn's Disease or 6-Point Mayo Score for Ulcerative Colitis; and Patient Satisfaction with the 'Health Promise' application.
  Arms: Nurse Follow-Up and Electronic Monitoring
Other: Post-Discharge Questionnaire — Patients will complete a web-based questionnaire at 30 days post-discharge. The questionnaire will capture information related to: Demographics, Patient Satisfaction as measured by the CACHE questionnaire; IBD related quality of life as measured by the IBDQ questionnaire; Disease activity as measured by PRO-2 scale for Crohn's Disease or 6-Point Mayo Score for Ulcerative Colitis.
  Arms: Minimal Intervention
Other: Standard of Care — Discharge summary detailing inpatient IBD admission; in addition to outpatient follow-up with a Gastroenterologist post-discharge

SUMMARY:
Patients with Inflammatory Bowel Disease (IBD) are frequently hospitalized, with an increased risk of repeat hospitalizations within the same calendar year. Given that hospital readmissions represent a significant burden to patients and the health care system, a standardised pathway for IBD patients discharged from the hospital can have a significant impact on reducing readmission rates, healthcare utilization and patient satisfaction. The primary aim of this study is to evaluate the effectiveness of an IBD post-discharge pathway, involving post-discharge nurse follow-up and electronic monitoring, in reducing IBD readmission rates.

DETAILED DESCRIPTION:
Background: Hospital readmission rates are a key issue in health policy as they place a large burden on the healthcare system. Readmissions are a preventable source of health care expenditure and in some cases, represent an opportunity for quality improvement. Lack of standardization in hospital discharge processes, and deficiencies in the transition of care after discharge, predispose patients to an increased risk of illness, hospital utilization and healthcare costs. Previously identified issues in discharge planning include timely transmission of discharge summaries to primary care providers and lack of communication between providers and patients with respect to discharge medications and follow-up appointments.

Rationale: Various post-discharge interventions have been effective in reducing hospital readmission rates and increasing patient satisfaction. However, in patients with flares of Inflammatory Bowel Disease (IBD), there is limited evidence to suggest which processes of care are protective against readmissions. IBD patients are frequently hospitalized, with over 22% of patients hospitalized within the first 2 years of diagnosis. Moreover, readmission rates are high in the IBD population, with over 20% of patients readmitted within the same calendar year of their initial hospitalization. Alongside increased healthcare expenditure, hospitalizations in the IBD population are associated with a number of nosocomial complications including venous thromboembolism and infection.

Specific Aim: The primary aim of this study is to determine whether standardized IBD post-discharge pathway, involving regular follow-up with an advanced practice nurse and electronic monitoring through a web-based application, decreases the risk of IBD readmissions when compared to the usual standard of care.

Study Design: All IBD inpatients with a diagnosis of Ulcerative Colitis (UC) or Crohn's Disease (CD) will be approached to participate in this parallel group randomized control trial. Patients randomized to the control arm will be discharged with the usual post-discharge standard of care. Patients randomized to the intervention arm will receive the usual post-discharge standard of care, in addition to organised follow-up with an advance practice nurse and electronic monitoring through a web-based application.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* IBD diagnosis of UC or CD
* Hospitalization for diagnosis or exacerbation of IBD

Exclusion Criteria:

* Inability to provide informed consent
* No internet access
* Death during hospitalization
* History of surgical management for IBD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Post-Discharge Readmission | Within 30 days of initial hospital discharge
  Occurrence of post-discharge readmissions will be recorded for all patients enrolled in the study. Post-discharge readmissions will be defined as any IBD readmission subsequent to the initial hospital admission where the patient was enrolled in the study. Post-discharge readmission rates will be compared between study arms.

SECONDARY OUTCOMES:
Post-Discharge Occurrence of Venous Thromboembolism | Within 30 days of initial hospital discharge
  Occurrence of post-discharge venous thromboembolism will be recorded for all patients enrolled in the study. Post-discharge occurrence of venous thromboembolism will be defined as any event of venous thromboembolism subsequent to the initial hospital admission where the patient was enrolled in the study. Post-discharge rates of venous thromboembolism will be compared between study arms.
Patient Satisfaction with Health Care in IBD | 30 days post-discharge
  Patient satisfaction with health care in IBD as measured by CACHE will be collected from all patients, through a web-based questionnaire administered at 30 days post-discharge of initial hospitalization; where patients were enrolled in the study. Mean scores for Patient Satisfaction with Health Care in IBD will be compared between study arms.
IBD related Quality of Life | 30 days post-discharge
  IBD related Quality of Life as measured by IBDQ will be collected from all patients, through a web-based questionnaire administered at 30 days post-discharge of initial hospitalization; where patients were enrolled in the study. Mean scores for IBD related Quality of Life will be compared between study arms.
Disease Activity | 30 days post-discharge
  Disease Activity as measured by PRO-2 for Crohn's Disease or 6-Point Mayo Score for Ulcerative Colitis will be collected from all patients, through a web-based questionnaire administered at 30 days post-discharge of initial hospitalization; where patients were enrolled in the study. Mean scores for disease activity will be compared between study arms.
Patient Satisfaction with 'Health Promise' | 30 days post-discharge
  Patient satisfaction with the 'Heath Promise' application will be collected from patients enrolled in the experimental arm, through a web-based questionnaire administered at 30 days post-discharge of initial hospitalization; where patients were enrolled in the study. Mean score for patient satisfaction the 'Health Promise' application will be interpreted.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Nguyen, MD, PhD, Principal Investigator — Mount Sinai Hospital, Canada
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Casellas F, Ginard D, Vera I, Torrejon A; GETECCU. Development and testing of a new instrument to measure patient satisfaction with health care in inflammatory bowel disease: the CACHE questionnaire. Inflamm Bowel Dis. 2013 Mar;19(3):559-68. doi: 10.1097/MIB.0b013e31827febd1. PMID 23429448
- [Background] Pallis AG, Mouzas IA, Vlachonikolis IG. The inflammatory bowel disease questionnaire: a review of its national validation studies. Inflamm Bowel Dis. 2004 May;10(3):261-9. doi: 10.1097/00054725-200405000-00014. PMID 15290922
- [Background] Hazratjee N, Agito M, Lopez R, Lashner B, Rizk MK. Hospital readmissions in patients with inflammatory bowel disease. Am J Gastroenterol. 2013 Jul;108(7):1024-32. doi: 10.1038/ajg.2012.343. PMID 23820989
- [Background] Vest JR, Gamm LD, Oxford BA, Gonzalez MI, Slawson KM. Determinants of preventable readmissions in the United States: a systematic review. Implement Sci. 2010 Nov 17;5:88. doi: 10.1186/1748-5908-5-88. PMID 21083908
- [Background] Makaryus AN, Friedman EA. Patients' understanding of their treatment plans and diagnosis at discharge. Mayo Clin Proc. 2005 Aug;80(8):991-4. doi: 10.4065/80.8.991. PMID 16092576
- [Background] Moore C, Wisnivesky J, Williams S, McGinn T. Medical errors related to discontinuity of care from an inpatient to an outpatient setting. J Gen Intern Med. 2003 Aug;18(8):646-51. doi: 10.1046/j.1525-1497.2003.20722.x. PMID 12911647
- [Background] Nguyen GC, Bollegala N, Chong CA. Factors associated with readmissions and outcomes of patients hospitalized for inflammatory bowel disease. Clin Gastroenterol Hepatol. 2014 Nov;12(11):1897-1904.e1. doi: 10.1016/j.cgh.2014.02.042. Epub 2014 Mar 26. PMID 24681074
- [Background] Bernstein CN, Nabalamba A. Hospitalization, surgery, and readmission rates of IBD in Canada: a population-based study. Am J Gastroenterol. 2006 Jan;101(1):110-8. doi: 10.1111/j.1572-0241.2006.00330.x. PMID 16405542
- [Background] Nguyen GC, Sam J. Rising prevalence of venous thromboembolism and its impact on mortality among hospitalized inflammatory bowel disease patients. Am J Gastroenterol. 2008 Sep;103(9):2272-80. doi: 10.1111/j.1572-0241.2008.02052.x. Epub 2008 Aug 5. PMID 18684186
- [Background] Nguyen GC, Kaplan GG, Harris ML, Brant SR. A national survey of the prevalence and impact of Clostridium difficile infection among hospitalized inflammatory bowel disease patients. Am J Gastroenterol. 2008 Jun;103(6):1443-50. doi: 10.1111/j.1572-0241.2007.01780.x. Epub 2008 May 29. PMID 18513271